CLINICAL TRIAL: NCT04899817
Title: Efficacy and Safety of Granisteron Versus Metoclopramide as Prophylaxis Antiemetic in Laparoscopic Cholecystectomy
Brief Title: Granisteron Versus Metoclopramide in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lyali Salah Dardeer, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Antiemetics in lab cholecystec
Record Dates: First submitted 2021-04-20; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Nausea and Vomiting, Postoperative
Keywords: Laparoscopic cholecystectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Granisetron

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group G (Active Comparator): will receive granisteron 1mg after induction of general anesthesia
  Interventions: Drug: Granisetron
- Group C (Placebo Comparator): Will receive metoclopramide 10 mg after induction of general anesthesia
  Interventions: Drug: Granisetron

INTERVENTIONS:
Drug: Granisetron — The drug is given after induction of general anesthesia
  Other Names: Granitryl

SUMMARY:
Study aims at comparing the effect of granisteron with that of metoclopramide in patients undergoing lab cholecystectomy

DETAILED DESCRIPTION:
Post operative nausea and vomitting is Avery common complication of laparoscopic surgery in that study we will compare between granisteron and metoclopramide as aprophlaxis against post operative nausea and vomitting

ELIGIBILITY:
Inclusion Criteria:

* both sexes Age between 18 and 60 years ASA1 2 3 Lap cholecystectomy under general anesthesia

Exclusion Criteria:

* patients refusal Pregnancy and breastfeeding Hepatic or renal disease ASA4 5 Allergy to the drug

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomitting | Every 2 hours for 12 hours
  Number of attacks of nausea and vomitting

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Esmail, Study Director — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt